CLINICAL TRIAL: NCT05366062
Title: Phase II Clinical Trial to Assess the Efficacy of ERC1671 to Treat Malignant Gliomas When Given in Combination With GM-CSF, Cyclophosphamide, Bevacizumab and Pembrolizumab in Patients Who Have Failed Prior Treatment With Radiation and Temozolomide
Brief Title: ERC1671 to Treat Malignant Gliomas When Given in Combination With GM-CSF, Cyclophosphamide, Bevacizumab and Pembrolizumab
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Epitopoietic Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERC1671PEM
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Glioma, Malignant
Keywords: ERC1671; GM-CSF; Cyclophosphamide; Bevacizumab; Pembrolizumab
MeSH Terms: conditions — Glioma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): This is a Treatment Protocol for patients with severe and immediately life-threatening GBM that had surgical resection and first line treatment with radiation therapy and temozolamide per current standard of care. Patients will be treated with recurring 28-day cycles of ERC1671, GM-CSF, Cyclophosphomide, Bevacizumab, and Pembrolizumab until progression of disease and at the discretion of the treating physician.
  Interventions: Drug: ERC1671; Drug: GM-CSF; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ERC1671 — ERC1671 is an autologous and allogeneic cells and lysates suspension generated from human glioblastoma (GBM) tumors harvested from patients undergoing surgery for glioblastoma. For each patient the treatment is composed of three allogeneic cells vaccine and lysates vaccine (ERC1671 A, B, C) plus from one autologous cells and lysate (ERC1671D).
Drug: GM-CSF — Sargramostim (Leukomax®, Leukine®); yeast-derived, recombinant human granulocyte-macrophage colony stimulating factor (rhu GM-CSF)
Drug: Cyclophosphamide — Cyclophosphamide is an alkylating agent, used for immunopotentiation. This drug is FDA approved and is being used off-label for the condition of hematopoietic stem cell transplant conditioning as an antineoplastic and immunosuppressant agent to modulate immunity.
Drug: Pembrolizumab — A therapeutic antibody that binds to and blocks PD-1 located on lymphocytes. The receptor is generally responsible for preventing the immune system from attacking the body's own tissues - it is an immune checkpoint inhibitor.
  Other Names: Keytruda

SUMMARY:
This is a treatment clinical trial to assess the efficacy of ERC1671 in combination with bevacizumab and pembrolizumab in patients with GBM that has progressed following treatment with radiation and temozolomide.

Patients will have surgery to collect the maximum amount of GBM tissue that can be reasonably collected. This tissue will be used to manufacturer ERC1671 for the patient.

The patients will receive ERC1671 in combination with GM-CSF and cyclophosphamide, in combination with bevacizumab and pembrolizumab.

DETAILED DESCRIPTION:
The treatment cycles will be 28 days long and follow the schedule below. There are 28 days (± 7 days) from surgery date to start of Cycle 1 day 1 to permit production of ERC-D vaccine:

The treatment will be repeated every 28-days until progression of disease, intolerance, or a decision by the physician and/or patient to withdraw from the treatment plan.

Efficacy will be evaluated as a foundation of Overall Survival reported at twelve months (OS12)

Safety will be evaluated, as a secondary objective, throughout the trial by the incidence of serious adverse events (AEs), physical examination findings, vital signs and clinical laboratory test results. SAEs will be graded for severity using NCI Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0.

Patients will undergo brain MRI as part of standard care before starting cycle 1 and every 8 weeks thereafter (+/- 7 days) until disease progression, and whenever progression is suspected based on clinical symptoms. Tumor response will be assessed using both the Macdonald and the iRANO response criteria for high-grade gliomas, which considers radiologic imaging, neurological status, and steroid dosing.

Whenever clinically appropriate, stereotactic biopsy or resection will be performed in accordance with standard of care for patients with progressive disease. To differentiate true progression from potentially toxic or therapeutic inflammatory responses presenting as radiographic or clinical changes, histologic verification of progression will be performed whenever feasible and appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of a recurrent/progressive WHO grade IV malignant gliomas (glioblastoma) and meet the following inclusion criteria:
* Age ≥18 years of age.
* KPS of ≥ 60%.
* Life expectancy > 12 weeks.
* First, second, third or fourth relapse of glioblastoma.
* Previous treatment for glioblastoma must include surgery (biopsy, partial resection, or full surgical resection), conventional radiation therapy and temozolomide (TMZ).
* MRI record must be obtained showing the MRI was done at least 4 weeks after any salvage surgery, and at least 12 weeks after radiation therapy, or at least 4 weeks after radiation for a new lesion outside the prior primary radiation field unless relapse is confirmed by tumor biopsy or new lesion outside of radiation field, or if there are two MRIs confirming progressive disease that are 8 weeks apart.
* If prior therapy with gamma knife or other focal high-dose radiation, must have subsequent histologic documentation of local relapse, or relapse with new lesion outside the irradiated field.
* Resolution of all chemotherapy or radiation-related toxicities ≤ CTCAE Grade severity, except for alopecia and hematologic toxicity. Patients taking temozolomide can start study treatment 23 days from the last temozolomide dose. For all other chemotherapy drugs, study treatment can start as long as all adverse events related to their prior treatment are no higher than Grade 1.
* Systemic corticosteroid therapy must be at a dose of ≤ 4 mg of dexamethasone or equivalent per day during the week prior to Day 1.
* Bi-dimensionally measurable disease (as per iRANO criteria).
* Patients must have normal organ and marrow function as defined below:
* Hemoglobin (Hbg) > 9g/dL,
* Leukocytes >1,500/mcL
* Absolute neutrophil count>1,000/mcL
* CD4 count > 300/mcl
* Platelets >125,000/mcL
* Serum bilirubin = 1.5 × upper limit of normal (ULN) or = 3 x ULN if Gilbert's disease is documented AST(SGOT) and ALT(SGPT)<2.5 x institutional upper limit of normal
* Serum creatinine < 1.5 mg/dl
* Signed informed consent approved by the Institutional Review Board;
* If sexually active, patients must agree to take contraceptive measures for the duration of the treatments.

Exclusion Criteria:

* Subjects unable to undergo an MRI with contrast
* Subjects able and willing to participate in an open and accruing ERC clinical trial
* Presence of diffuse leptomeningeal disease
* History, presence, or suspicion of metastatic disease
* Administration of immunosuppressive drugs less than 2 weeks prior to first dose of ERC1671 except dexamethasone for cerebral edema as detailed above;
* Known contraindication or hypersensitivity to any component of bevacizumab.
* Evidence of recent hemorrhage on screening MRI of the brain with the following exceptions: presence of hemosiderin; resolving hemorrhagic changes related to surgery; presence of punctate hemorrhage in the tumor.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1.
* Evidence of bleeding diathesis or coagulopathy as documented by an elevated PT, PTT or bleeding time and clinically significant;
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to Day 1.
* Urine protein: creatinine ratio 1.0 at screening;
* Anticipation of need for major surgical procedure during the course of the study.
* Serious non-healing wound, ulcer, or bone fracture.
* Active infection requiring treatment, known immunosuppressive disease, active systemic autoimmune diseases such as lupus, receipt of systemic immunosuppressive therapy, human immunodeficiency virus (HIV) infection, Hepatitis B or Hepatitis C.
* Uncontrolled hypertension, blood pressure of > 150 mmHg systolic and > 100 mmHg diastolic, or history of hypertensive encephalopathy. Subjects with any known uncontrolled inter-current illness including ongoing or active infection, symptomatic congestive heart failure (NYHA Gr.2 or >), myocardial infarction, unstable angina pectoris within the past 12 months
* Stroke, transient ischemic attack, unstable angina, myocardial infarction or congestive heart failure (New York Heart Association Grade II or greater) within the past 12 months. Unstable or severe intercurrent medical conditions, chronic renal disease, or uncontrolled diabetes mellitus.
* Women who are pregnant or lactating. All female patients with reproductive potential must have a negative pregnancy test prior to Day 1 and agree to use reliable contraception whilst study participant.
* Men refusing to exercise a reliable form of contraception.
* History of any malignancy (other than glioblastoma) during the last three years except non-melanoma skin cancer, in situ cervical cancer, treated superficial bladder cancer or cured, early-stage prostate cancer in a patient with Prostate Surface Antigen (PSA) level <ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival at 12 months | 12 months
  Overall Survival at 12 months as assessed per iRANO Criteria.

SECONDARY OUTCOMES:
Progression-free survival | 12 Months
  Dates from date of first injection of vaccine.
Radiographic Response | 12 Months
  Radiographic Response, categorized per iRANO Criteria.
Number of participants with Adverse Events [Safety and Tolerability] | 12 months
  As indicated by the number and rate of adverse events, categorized by the CTCAE v. 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Bumrungrad International Hospital, Bangkok, Vadhana, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barker FG 2nd, Chang SM, Gutin PH, Malec MK, McDermott MW, Prados MD, Wilson CB. Survival and functional status after resection of recurrent glioblastoma multiforme. Neurosurgery. 1998 Apr;42(4):709-20; discussion 720-3. doi: 10.1097/00006123-199804000-00013. PMID 9574634
- [Background] Ben-Efraim S. Immunomodulating anticancer alkylating drugs: targets and mechanisms of activity. Curr Drug Targets. 2001 Jun;2(2):197-212. doi: 10.2174/1389450013348597. PMID 11469719
- [Background] BLOOM WH, CARSTAIRS KC, CROMPTON MR, McKISSOCK W. Autologous glioma transplantation. Lancet. 1960 Jul 9;2(7141):77-8. doi: 10.1016/s0140-6736(60)91219-8. No abstract available. PMID 13801625
- [Background] Bowles AP Jr, Perkins E. Long-term remission of malignant brain tumors after intracranial infection: a report of four cases. Neurosurgery. 1999 Mar;44(3):636-42; discussion 642-3. doi: 10.1097/00006123-199903000-00110. PMID 10069601
- [Background] Brem S, Cotran R, Folkman J. Tumor angiogenesis: a quantitative method for histologic grading. J Natl Cancer Inst. 1972 Feb;48(2):347-56. No abstract available. PMID 4347034
- [Background] Bystryn JC, Rigel D, Friedman RJ, Kopf A. Prognostic significance of hypopigmentation in malignant melanoma. Arch Dermatol. 1987 Aug;123(8):1053-5. PMID 3631983
- [Background] Clarke JL, Ennis MM, Yung WK, Chang SM, Wen PY, Cloughesy TF, Deangelis LM, Robins HI, Lieberman FS, Fine HA, Abrey L, Gilbert MR, Mehta M, Kuhn JG, Aldape KD, Lamborn KR, Prados MD; North American Brain Tumor Consortium. Is surgery at progression a prognostic marker for improved 6-month progression-free survival or overall survival for patients with recurrent glioblastoma? Neuro Oncol. 2011 Oct;13(10):1118-24. doi: 10.1093/neuonc/nor110. Epub 2011 Aug 2. PMID 21813511
- [Background] Coley WB. The treatment of malignant tumors by repeated inoculations of erysipelas. With a report of ten original cases. 1893. Clin Orthop Relat Res. 1991 Jan;(262):3-11. No abstract available. PMID 1984929
- [Background] Crane CH, Ellis LM, Abbruzzese JL, Amos C, Xiong HQ, Ho L, Evans DB, Tamm EP, Ng C, Pisters PW, Charnsangavej C, Delclos ME, O'Reilly M, Lee JE, Wolff RA. Phase I trial evaluating the safety of bevacizumab with concurrent radiotherapy and capecitabine in locally advanced pancreatic cancer. J Clin Oncol. 2006 Mar 1;24(7):1145-51. doi: 10.1200/JCO.2005.03.6780. PMID 16505434
- [Background] D'Adamo DR, Anderson SE, Albritton K, Yamada J, Riedel E, Scheu K, Schwartz GK, Chen H, Maki RG. Phase II study of doxorubicin and bevacizumab for patients with metastatic soft-tissue sarcomas. J Clin Oncol. 2005 Oct 1;23(28):7135-42. doi: 10.1200/JCO.2005.16.139. PMID 16192597
- [Background] Dang Y, Wagner WM, Gad E, Rastetter L, Berger CM, Holt GE, Disis ML. Dendritic cell-activating vaccine adjuvants differ in the ability to elicit antitumor immunity due to an adjuvant-specific induction of immunosuppressive cells. Clin Cancer Res. 2012 Jun 1;18(11):3122-31. doi: 10.1158/1078-0432.CCR-12-0113. Epub 2012 Apr 17. PMID 22510348
- [Background] Deorah S, Lynch CF, Sibenaller ZA, Ryken TC. Trends in brain cancer incidence and survival in the United States: Surveillance, Epidemiology, and End Results Program, 1973 to 2001. Neurosurg Focus. 2006 Apr 15;20(4):E1. doi: 10.3171/foc.2006.20.4.E1. PMID 16709014
- [Background] Emens LA. GM-CSF-secreting vaccines for solid tumors. Curr Opin Investig Drugs. 2009 Dec;10(12):1315-24. PMID 19943203
- [Result] Ammirati M, Galicich JH, Arbit E, Liao Y. Reoperation in the treatment of recurrent intracranial malignant gliomas. Neurosurgery. 1987 Nov;21(5):607-14. doi: 10.1227/00006123-198711000-00001. PMID 2827051